CLINICAL TRIAL: NCT00866268
Title: "Low Versus High Pressure Suction Drainage After Total Knee Arthroplasty: a Double Blind Randomized Controlled Trial"
Brief Title: Low Versus High Pressure Suction Drainage After Total Knee Arthroplasty
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Rafa Calvo Oyón, Hospital de la Santa Creu i Sant Pau
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DRENAJE50MMHG/1
Record Dates: First submitted 2009-03-19; First posted 2009-03-20 (Estimated); Last update posted 2009-03-20 (Estimated); Status verified 2009-03

CONDITIONS: Total Knee Arthroplasty
Keywords: Blood loss; Total knee arthroplasty; Adults; Drain; Drainage system
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low suction drainage (Experimental): In the experimental group the drainage catheter was connected to a modified DRENOFAST® system. This system consisted of a sterile plastic bottle with a holding capacity of 600 mL of fluid and a negative pressure of 700mmHg. It was hermetically closed and had two connections. The DRENOFAST® modification consisted of establishing an open connection between the bottle and a wall vacuum source (normally used to administer oxygen) placed next to the patient's bed. The 50 mmHg constant negative pressure of the bottle was maintained by the wall vacuum source and verified by flow meter.
  Interventions: Device: low pressure suction drainage
- High suction drainage (Active Comparator): The standard DRENOFAST® system was used in the control group, and the initial negative pressure was 700 mmHg.
  Interventions: Device: High pressure suction drainage

INTERVENTIONS:
Device: low pressure suction drainage — In the experimental group the drainage catheter was connected to a modified DRENOFAST® system. This system consisted of a sterile plastic bottle with a holding capacity of 600 mL of fluid and a negative pressure of 700mmHg. It was hermetically closed and had two connections. The DRENOFAST® modification consisted of establishing an open connection between the bottle and a wall vacuum source (normally used to administer oxygen) placed next to the patient's bed. The 50 mmHg constant negative pressure of the bottle was maintained by the wall vacuum source and verified by flow meter. Duration: Drains were removed after bleeding had ceased (48-72h).
  Other Names: DRENOFAST® modified
  Arms: Low suction drainage
Device: High pressure suction drainage — In order to mask the type of intervention from the patient and the investigators, both drainage systems had two drain catheters. One catheter allowed the blood to flow from the wound to the bottle. The second catheter connected the bottle to the vacuum source. In the experimental arm the second catheter was open, while in the control group it was closed. So that the system used could not be distinguished, the connection of the second catheter to the bottle was covered with opaque adhesive tape.Drains were removed after bleeding had ceased.
  Other Names: DRENOFAST® system
  Arms: High suction drainage

SUMMARY:
Principal hypothesis:

A low suction drainage (-50 mmHg) reduce a 25% the blood loss with respect a standard closed drainage (-700 mmHg) following total knee arthroplasty.

DETAILED DESCRIPTION:
Secondary's hypothesis:

* It don't expect differences in:

  1. Incidence of hematomas
  2. Incidence in surgery wound infection
  3. Time of immobilization
  4. Duration of hospitalization
* The low suction drainage (-50 mmHg) will be more cost-effective than the standard closed drainage (-700 mmHg)

ELIGIBILITY:
Inclusion Criteria:

* Adult knee replacement patients who agreed to participate in the study

Exclusion Criteria:

* People that not accomplished the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2006-05; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
total post-surgical blood loss (mL) | from the moment after surgery until drainage catheter removal

SECONDARY OUTCOMES:
blood loss (mL) in the recovery unit | 24-48 h
Blood loss in the ward | 5-10 days
need for a blood transfusion according to the surgeon's criteria | 10 days
number of blood units required for transfusion | 10 Days
post-surgical pain (using a 100mm visual analogue scale) | 10 days
incidence of hematomas | 10 days
infections | 10 days
suture dehiscence | 10 days
re-intervention due to complications in the surgical wound | 10 dasy
venous thrombosis | 10 days
hypotension | 10 days
mortality | 10 days
adverse reactions | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Calvo Rafael, Rn, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (2):
- Spain (2):
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia
  - Orthopedic and Traumatology Service. Hospital de la Santa Creu i Sant Pau., Barcelona, Catalonia